CLINICAL TRIAL: NCT00229281
Title: Short Term Group Therapy for Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3680-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders | interventions — Psychotherapy, Group

INTERVENTIONS:
Behavioral: Group therapy

SUMMARY:
Assessing Anxiety in patient suffering from anxiety disorders (NOT OCD or PTSD)before and after group therapy

ELIGIBILITY:
Inclusion Criteria:

* Anxiety disorder (other than OCD or PTSD)
* Eligibility to participate in group therapy

Exclusion Criteria:

* OCD
* PTSD
* Suicidal thoughts
* Psychotic state
* Severe hostile personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel